CLINICAL TRIAL: NCT02695199
Title: Comparison Between Laparoscopic Doppler Ultrasound Assisted Laparoscopic Varicocelectomy and Microscopic Subinguinal Varicocelectomy
Brief Title: Doppler Ultrasound Assisted Varicocelectomy Improve Sperm Qualities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49557309-6
Record Dates: First submitted 2016-01-21; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-01

CONDITIONS: Varicocele
Keywords: Doppler Ultrasound; Laparoscopic; Microscopic Subinguinal Varicocelectomy
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic varicocelectomy (Experimental): laparoscopic Doppler ultrasound assisted laparoscopic varicocelectomy group
  Interventions: Procedure: Laparoscopic varicocelectomy
- microscopic varicocelectomy (Sham Comparator): conventional Microscopic Subinguinal varicocelectomy group
  Interventions: Procedure: Microscopic Subinguinal varicocelectomy

INTERVENTIONS:
Procedure: Laparoscopic varicocelectomy — Traditional laparoscopic varicocelectomy assisted by laparoscopic Doppler ultrasound
  Other Names: Laparoscopic varicocelectomy assisted by Doppler ultrasound
  Arms: laparoscopic varicocelectomy
Procedure: Microscopic Subinguinal varicocelectomy — Infertile patients with clinically palpable varicoceles were selected to receive microscopic Subinguinal varicocelectomy
  Other Names: Traditional microscopic Subinguinal varicocelectomy
  Arms: microscopic varicocelectomy

SUMMARY:
To evaluate the benefits of laparoscopic Doppler ultrasound (LDU) assisted laparoscopic varicocelectomy (LV) and compare the surgical outcomes and complications between LDU assisted LV (LDU-LV) and microscopic subinguinal varicocelectomy for infertile patients with varicoceles.

DETAILED DESCRIPTION:
To compare the surgical outcomes such as semen parameters and the pregnancy rate and complications like postoperative varicocele recurrence and hydrocele between laparoscopic Doppler ultrasound assisted laparoscopic varicocelectomy and conventional microscopic subinguinal for infertile patients with varicoceles. To examine the microanatomy of the spermatic cord within suprainguinal portion.

ELIGIBILITY:
Inclusion Criteria:

1. 20-39 years old who had infertility for more than 1 year and had clinical palpable varicoceles;
2. impaired semen quality including sperm concentration <15 million/ml or total motility <40% or progressively motile < 32% (a+b), the 5th edited World Health Organization criteria was referred;
3. with normal level of serum hormones including follicle stimulating hormone, luteinizing hormone, Thyroid hormones and prolactin;
4. patient's spouse was healthy in reproduction.

Exclusion Criteria:

1. with subclinical varicocele, recurrent varicoceles;
2. normal semen analyses;
3. other reasons of infertility than varicoceles;
4. refusing to enter randomization;
5. female partner older than 35 years;
6. with abnormal level of serum hormones;
7. female factor infertility;
8. with significant surgical diseases, congenital diseases or endocrine diseases.

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | The pregnancy rate was calculated at 1 year of follow-up

SECONDARY OUTCOMES:
semen quality assessment | semen quality assessment were checked at 3, 6 and 12 months after surgery.
  Routine sperm quality check including Count，Morphology and Motility using both the conventional manual method and computer assisted sperm analysis (CASA) systems.
postoperative complications | postoperative complications at 3, 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhen Yuan, MD, Study Director — Second hospital of Shandong University
Locations (1):
- Second Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided